CLINICAL TRIAL: NCT02681549
Title: A Phase 2 Trial of Pembrolizumab Plus Bevacizumab in Patients With Metastatic Melanoma or Non-small Cell Lung Cancer With Untreated Brain Metastases
Brief Title: Pembrolizumab Plus Bevacizumab for Treatment of Brain Metastases in Metastatic Melanoma or Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Harriet Kluger, Principal Investigator, Yale University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1512016953; 1511MEL007 (Other Grant/Funding Number: Merck Sharp & Dohme LLC); 1R01CA269286-01A1 (NIH)
Record Dates: First submitted 2016-02-09; First posted 2016-02-12 (Estimated); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Melanoma; Non-small Cell Lung Cancer; Brain Metastasis
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — pembrolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Untreated brain metastases from melanoma (Experimental): pembrolizumab plus bevacizumab
  Interventions: Drug: Pembrolizumab plus Bevacizumab
- Untreated brain metastases from NSCLC (Experimental): pembrolizumab plus bevacizumab
  Interventions: Drug: Pembrolizumab plus Bevacizumab

INTERVENTIONS:
Drug: Pembrolizumab plus Bevacizumab — Pembrolizumab will be administered on day 1 of every cycle until disease progression or withdrawal from study. Bevacizumab will be administered in addition to pembrolizumab on day 1 of cycles 1, 2, 3, and 4 (or alternative cycles if bevacizumab is held during these cycles). Three weeks constitutes one cycle.

SUMMARY:
The purpose of this phase 2 trial is to study the activity of pembrolizumab in combination with bevacizumab in patients with untreated brain metastases from melanoma or NSCLC to determine activity and safety of the drug combination. Furthermore, in patients who undergo resection of biopsy of a brain metastasis, we will evaluate biomarkers predictive of treatment benefit, and will also conduct correlative biomarker studies on extra-cerebral specimens in all patients in whom a systemic biopsy is feasible or in archival tumor tissue when available.

A total of 53 eligible patients will be enrolled on this trial (40 with melanoma and 13 with NSCLC). Individual cohorts of the study can be stopped if insufficient activity is observed in the first stage of that cohort. The study will accrue for approximately 84 months, and will be open for approximately 12 additional months as patients on study are being followed.

ELIGIBILITY:
Major Inclusion Criteria:

1. Biopsy proven metastatic melanoma or non-squamous NSCLC with at least one untreated brain metastasis that is at least 5 mm AND twice the MRI slice thickness, but less than 20 mm, which is asymptomatic and not requiring immediate local therapy or steroids.
2. Patients who have had prior resection or biopsy of a CNS metastasis will be required to provide a paraffin embedded specimen from tumor taken at the time of surgery, if available.
3. Patients will be required to undergo biopsy or submit archival tumor tissue from a systemic site of disease for correlative studies. When not feasible, this requirement can be waived after discussion with the principal investigators.
4. PD-L1 expression in tumor tissue from any site determined by the Dako 22C3 assay is required for patients with NSCLC.
5. Adequate organ function.
6. ECOG performance status < 2.
7. Any number of previous treatments with the exception of previous inhibitors of PD-1 or PD-L1.
8. Life expectancy of at least 3 months.
9. Understanding and willingness to consent.
10. A history of radiotherapy for brain metastases is allowed, but any lesion present at the time of WBRT or included in the stereotactic radiotherapy field will NOT be considered evaluable unless documented to have progressed since treatment.

Overall Inclusion Criteria:

1. Biopsy proven metastatic melanoma or non-squamous NSCLC with at least one untreated cerebral metastasis that is at least 5 mm AND twice the MRI slice thickness, but less than 20 mm, that is asymptomatic and does not require local therapy at the time of enrollment ("clinically evaluable lesion(s)"). An untreated brain metastasis is defined as a lesion not present at the time of whole brain radiation therapy or included in a stereotactic radiotherapy field (or within 2mm of a treated lesion), or any lesion that is new or unequivocally progressing since prior radiation therapy.
2. ECOG performance status < 2
3. Any number of previous treatments with the exception of previous inhibitors of PD-1, PD-L1, or PD-L2. Other prior systemic therapies must have been administered at least 2 weeks before administration of pembrolizumab; the exception to this is ipilimumab which must have been administered at least 4 weeks prior to the start of pembrolizumab. Patients are not required to have had prior systemic therapy.
4. Life expectancy of at least 3 months
5. A history of previously treated brain metastases is allowed, provided that at least 7 days have lapsed between radiation and initiation of pembrolizumab. Any brain metastasis ≥ 20mm or causing symptoms must be treated with local therapy (i.e. radiation or surgical resection, as clinically appropriate) prior to study enrollment. Any lesion present at the time of WBRT or included in the stereotactic radiotherapy field (or within 2mm of the treated lesion) will NOT be considered evaluable unless it is new or documented to have progressed since treatment.
6. PD-L1 expression >1% in tumor tissue from any site is required for patients with NSCLC. Tumor tissue can be archival if no intercurrent systemic therapy was administered, however if no archival tissue is available or if intercurrent systemic therapy was administered, then a biopsy must be obtained for PD-L1 testing. PD-L1 expression must be obtained using the Dako 22C3 assay in a CLIA-certified laboratory. PD-L1 expression is not required for patients with melanoma.
7. All patients are required to submit a tumor specimen for analysis (brain or extra-cerebral). A formalin-fixed paraffin-embedded (FFPE) tissue block, or a 4mm punch from an FFPE block must be submitted. If it is not possible to safely obtain a biopsy due to anatomic location of tumors, and no prior tissue is available, this requirement may be waived upon discussion with the study PI or co-PI.
8. Patients must have normal organ and marrow function (as defined in the protocol) at the time of screening.
9. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
11. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Major Exclusion Criteria:

1. Symptomatic brain metastases at the time of initiation of systemic therapy.
2. Other systemic therapy within 14 days of initiation of study drug.
3. Use of corticosteroids to control CNS symptoms. Low-dose steroid use (≤10 mg of prednisone or equivalent) is allowed.
4. Presence of leptomeningeal disease.
5. Presence of active autoimmune disease. Autoimmune thyroid disease will be allowed if thyroid function is within normal range.

Overall Exclusion Criteria:

1. Symptomatic brain metastases. Any neurologic symptoms present must have resolved with local therapy by the time of administration of study drug.
2. Patients with brain metastases for whom complete surgical resection is clinically appropriate.
3. Patients with lung cancer with squamous histology.
4. Has had prior chemotherapy or targeted small molecule therapy within 2 weeks prior to start of treatment or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Previous radiation to extracranial sites may be completed at any time prior to initiation of pembrolizumab.

   1. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
   2. Note: Toxicity that has not recovered to ≤ Grade 1 is allowed if it meets the inclusion requirements for laboratory parameters.
5. Has had prior treatment with any other anti-PD-1 or PD-L1 or PD-L2 agent.
6. The use of corticosteroids to control cerebral edema or treat neurologic symptoms will not be allowed, and patients who previously required corticosteroids for symptom control must be off steroids for at least 1 week prior to treatment on day 1 of cycle 1. Low-dose steroid use (≤10 mg of prednisone or equivalent) as corticosteroid replacement therapy is allowed
7. Has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
8. Presence of leptomeningeal disease
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Pregnancy or breast feeding. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pembrolizumab, breastfeeding must be discontinued if the mother is treated with pembrolizumab.
11. Patients may not be receiving any other investigational agents and may not have participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
12. Either a concurrent condition (including medical illness, such as active infection requiring treatment with intravenous antibiotics or the presence of laboratory abnormalities) or history of a prior condition that places the patient at unacceptable risk if he/she were treated with the study drug or a medical condition that confounds the ability to interpret data from the study.
13. Concurrent, active malignancies in addition to those being studied (other than cutaneous squamous cell carcinoma or basal cell carcinoma)
14. Patients with active hemoptysis.
15. Any contraindication to MRI (i.e. patients with pacemakers or other metal implanted medical devices). An MRI safety questionnaire is required prior to MR imaging.
16. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
17. Has a known Human Immunodeficiency Virus (HIV), Hepatitis B (HBV), or Hepatitis C (HCV) infection.
18. Has received a live vaccine within 30 days prior to the first dose of trial treatment.
19. Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure > 100 mmHg). Anti-hypertensive therapy to achieve these parameters is allowable.
20. History of myocardial infarction or unstable angina within 3 months prior to Cycle 1, Day 1
21. History of stroke or transient ischemic attack within 3 months prior to Cycle 1, Day 1
22. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Cycle 1, Day 1
23. Evidence of bleeding diathesis or clinically significant coagulopathy (in the absence of therapeutic anticoagulation). Any history of significant bleeding or thrombosis should be discussed the study PIs.
24. Current or recent (within 10 calendar days prior to Cycle 1, Day 1) use of dipyramidole, ticlopidine, clopidogrel, or cilostazol
25. Warfarin is not permitted. Prophylactic or therapeutic use of low molecular-weight heparin (e.g., enoxaparin) or direct thrombin inhibitors are permitted.
26. History of abdominal or tracheoesophageal fistula or gastrointestinal perforation within 6 months prior to Cycle 1, Day 1
27. Serious, non-healing or dehiscing wound
28. Proteinuria > 2.0 g of protein in a 24-hour urine collection. All patients with 2 protein on dipstick urinalysis at baseline must undergo a 24-hour urine collection for protein.
29. Has a history of (non-infectious) pneumonitis that required steroids, current pneumonitis or evidence of interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriett Kluger, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weiss SA, Djureinovic D, Wei W, Tran T, Austin M, Markowitz J, Eroglu Z, Khushalani NI, Hegde U, Cohen J, Sznol M, Anderson G, Johnson B, Piteo C, Mahajan A, Adeniran A, Jilaveanu L, Goldberg S, Chiang V, Forsyth P, Kluger HM. Phase II Trial of Pembrolizumab in Combination With Bevacizumab for Untreated Melanoma Brain Metastases. J Clin Oncol. 2025 May 10;43(14):1685-1694. doi: 10.1200/JCO-24-02219. Epub 2025 Mar 6. PMID 40048689

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Untreated Brain Metastases From Melanoma | Untreated Brain Metastases From NSCLC
Started | 37 | 4
Completed | 37 | 2
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Untreated Brain Metastases From Melanoma | Untreated Brain Metastases From NSCLC | Total
Number analyzed (Participants) | 37 | 4 | 41
Age, Continuous [Median (Full Range); unit: years] | 66 [32 to 88] | 67 [66 to 82] | 66 [32 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 27 | 1 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 34 | 3 | 37
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 36 | 3 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 37 | 5 | 42
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: units on a scale] — ECOG Performance Status (PS) is a scale that measures how a patient's cancer affects their daily life and ability to function. 0: Normal activity, 1: Some symptoms, but still mostly ambulatory.
  units on a scale
    0 | 25 | 1 | 26
    1 | 12 | 4 | 16
Mutation Status [Number; unit: participants] — Number of participants with each of the mutations listed below. Population: This measure does not apply to NSCLC group.
  participants
    BRAF WT: number analyzed (Participants) | 37 | 0 | 37
    BRAF WT | 19 |  | 19
    BRAF Mutant: number analyzed (Participants) | 37 | 0 | 37
    BRAF Mutant | 16 |  | 16
    V600E: number analyzed (Participants) | 37 | 0 | 37
    V600E | 9 |  | 9
    V600K: number analyzed (Participants) | 37 | 0 | 37
    V600K | 6 |  | 6
    Unknown V600 type: number analyzed (Participants) | 37 | 0 | 37
    Unknown V600 type | 1 |  | 1
    NRAS Mutant: number analyzed (Participants) | 37 | 0 | 37
    NRAS Mutant | 4 |  | 4
    Unknown Mutation Status: number analyzed (Participants) | 37 | 0 | 37
    Unknown Mutation Status | 2 |  | 2
Serum lactate dehydrogenase [Count of Participants; unit: Participants] — Population: This measure does not apply to NSCLC group.
  Participants
    Normal levels: number analyzed (Participants) | 37 | 0 | 37
    Normal levels | 25 | 0 | 25
    Elevated levels: number analyzed (Participants) | 37 | 0 | 37
    Elevated levels | 12 | 0 | 12
Number of intracranial target lesions [Count of Participants; unit: Participants]
  1-2 | 23 | 4 | 27
  3-5 | 14 | 0 | 14
Presence of extracranial metastases [Count of Participants; unit: Participants]
  Yes | 32 | 4 | 36
  No | 5 | 0 | 5
Prior systemic therapy [Count of Participants; unit: Participants]
  Yes | 7 | 0 | 7
  No | 30 | 4 | 34
Prior local therapy for MBM [Count of Participants; unit: Participants]
  Yes | 19 | 2 | 21
  No | 18 | 3 | 21

OUTCOME MEASURES:

1. Primary Outcome: Brain Metastasis Response Rate (BMRR)
Description: Brain metastasis response rate (BMRR) using modified RECIST (mRECIST) criteria
Time Frame: up to 2 years from start of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Untreated Brain Metastases From Melanoma | Untreated Brain Metastases From NSCLC
Number analyzed (Participants) | 37 | 4
percentage of participants | 54.1 | 75

2. Secondary Outcome: Steroid Use
Description: Number of patients using steroids to control of cerebral edema for greater than 96 hours
Time Frame: up to 2 years from start of treatment
Population: At time of analysis it was found that data reported by participants was incorrect and could not be used.
Measure: Count of Participants; unit: Participants
Arm/Group | Untreated Brain Metastases From Melanoma | Untreated Brain Metastases From NSCLC
Number analyzed (Participants) | 37 | 4
Participants | 3 | 1

3. Secondary Outcome: Overall Response Rate (ORR)
Description: best overall response rate (ORR) by mRECIST criteria in the brain or RECIST criteria in the body
Time Frame: up to 2 years from start of treatment
Population: Denominator for extracranial response is 32 because 5 patients did not have extracranial metastases at baseline
Measure: Number; unit: percentage of participants
Arm/Group | Untreated Brain Metastases From Melanoma | Untreated Brain Metastases From NSCLC
Number analyzed (Participants) | 37 | 4
percentage of participants
  Intracranial | 54.1 | 75
  Extracranial: number analyzed (Participants) | 32 | 4
  Extracranial | 56.3 | 75

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival by mRECIST criteria in the brain or RECIST criteria in the body
Time Frame: up to 9 years from start of treatment or to disease progression
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Untreated Brain Metastases From Melanoma | Untreated Brain Metastases From NSCLC
Number analyzed (Participants) | 37 | 4
years
  Median intracranial PFS | 2.2 [0.41 to NA] — Due to small sample size and censoring, upper limit could not be calculated | NA [NA to NA] — Due to small sample size and censoring, PFS could not be calculated
  Median overall PFS | 1.2 [0.23 to NA] — Due to small sample size and censoring, upper limit could not be calculated | NA [NA to NA] — Due to small sample size and censoring, PFS could not be calculated

5. Secondary Outcome: Safety and Toxicity of Combination Pembrolizumab and Bevacizumab Assessed Using Common Terminology Criteria for Adverse Events v. 4.
Description: Number of participants that experienced at least 1 treatment related adverse event.
Time Frame: up to 2 years from start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Untreated Brain Metastases From Melanoma | Untreated Brain Metastases From NSCLC
Number analyzed (Participants) | 37 | 4
Participants | 32 | 3

6. Other Pre Specified Outcome: PD-L1 Expression and Other Potential Predictive Biomarkers in CNS, Tumors and Blood, Correlated With Response to Treatment
Time Frame: 2 years from start of trial
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 2 years from the start of treatment
Arm/Group | Untreated Brain Metastases From Melanoma | Untreated Brain Metastases From NSCLC
All-Cause Mortality (participants affected / at risk) | 1/37 | 0/5
Serious Adverse Events (participants affected / at risk) | 4/37 | 1/5
Other Adverse Events (participants affected / at risk) | 27/37 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Untreated Brain Metastases From Melanoma (N=37) | Untreated Brain Metastases From NSCLC (N=5)
Investigations - Other, specify (Investigations) | 2 | 0 — Increased alanine aminotransferase (ALT)
Hypophysitis (Endocrine disorders) | 1 | 0
Wound dehiscence and infection (Vascular disorders) | 1 | 0
Pericardial tamponade (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Untreated Brain Metastases From Melanoma (N=37) | Untreated Brain Metastases From NSCLC (N=5)
Fatigue (General disorders) | 9 | 1
Rash (Skin and subcutaneous tissue disorders) | 8 | 0
Arthralgias (Musculoskeletal and connective tissue disorders) | 7 | 0
Investigations - Other, specify (Investigations) | 2 | 0 — Increased alanine aminotransferase (ALT)
Hypothyroidism (Endocrine disorders) | 4 | 0
Investigations - Other, specify (Investigations) | 5 | 0 — Increased aspartate aminotransferase (AST)
Pruritis (Skin and subcutaneous tissue disorders) | 3 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 3 | 0
Investigations - Other, specify (Investigations) | 2 | 0 — Increased bilirubin
Diarrhea (Gastrointestinal disorders) | 2 | 0
Investigations - Other, specify (Investigations) | 2 | 0 — Increased creatinine
Mucositis (Gastrointestinal disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 2
Dry eyes (Eye disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Investigations - Other, specify (Investigations) | 1 | 0 — Cardiac troponin increase
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Gingival bleed (General disorders) | 1 | 0
Microscopic diverticular perforation (Gastrointestinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 2
Headache (Nervous system disorders) | 15 | 0
Motor neuropathy (Nervous system disorders) | 3 | 0
Sensory neuropathy (Nervous system disorders) | 3 | 0
Stroke (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Encephalitis (Nervous system disorders) | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0 — Tingling of Arms and Legs
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 — C Diff Infection
Fall (Injury, poisoning and procedural complications) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Pain- Abdominal (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 0
Parainfluenza (Infections and infestations) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 1 | 0
Intracranial Hemorrage (Nervous system disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Thromboembolic Event (Vascular disorders) | 2 | 0
Ventriculitis (Cardiac disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1 — Black tarry stools
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 1 — SWEATS, INTERMITTENT
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 2 — Diverticulitis
Floaters (Eye disorders) | 0 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 1 — Taste Alteration
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1 — Deep vein thrombosis
Constipation (Gastrointestinal disorders) | 0 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 1 — Pain - Left Rib Intermittent
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 1 — Pain-Lower abdominal (heaviness feeling)
Hypothyroidism (Endocrine disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Hemoplysis- Intermittent

LIMITATIONS AND CAVEATS:
At time of analysis it was found that data reported by participants for the Steroid Use outcome was incorrect and therefore unreliable and could not be used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT02681549/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-09): https://cdn.clinicaltrials.gov/large-docs/49/NCT02681549/ICF_001.pdf